CLINICAL TRIAL: NCT05216185
Title: The Assessment of Bone Health in a Clinical Setting
Status: Not yet recruiting | Type: Observational
Sponsor: Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: RL1 842
Record Dates: First submitted 2022-01-17; First posted 2022-01-31 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-01

CONDITIONS: Case Series/Case Note Review

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will use data already obtained through the metabolic clinical service to improve diagnosis and management of our patients.

DETAILED DESCRIPTION:
Patients are referred for assessment of their bone health routinely have a bone density (BD) scan (DXA) and many also have a bone marker (BM) measurement, either NTx ( breakdown product of bone) or PINP ( formation product of bone). Patients diagnosed with osteoporosis are usually treated with a bisphosphonate drug which can halt or at least decrease the rate of bone loss.

BMs are measured pre- and post -treatment to assess adherence and effectiveness of treatment. BD measured by DXA is also used for this but in clinical practice is not recommended at intervals of less than 2 years. BMs show a much earlier clinical meaningful change - typically 2-6 months, vs BD -typically 2 years, thereby aiding swift knowledge of response or lack of response to treatment.

Although DXA remains the gold standard for initial assessment of bone health by measuring BD, BMs have an increasing role to play in patient follow up.

We propose to interrogate available data to explore whether utilizing BMs can provide monitoring information up to 5 years post-treatment thereby increasing the follow up time of the next DXA scan. This would ensure patients are not being subjected to scans using x-rays unduly and that a DXA scan is only performed when clinically needed. Additionally we want to investigate if BM levels pre-treatment reflect the response to treatment of the marker and BD, prediction of BM levels from age, fracture history, treatment, and does site of fracture affect BM and BD.

Previous work by other investigators has covered some of this ground but has not come up with definitive answers.

The study is expected to take 5 years and will not involve additional investigations compared to standard care.

ELIGIBILITY:
Inclusion Criteria: All patients on database -

Exclusion Criteria: Not recruiting

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on database
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Use of Bone markers as a surrogate for Bone mineral density | 5 years
  The study aims to use data already obtained through the clinical service to improve diagnosis and management of our patients. We aim to assess whether bone markers can be utilised more effectivley, thereby reducing the frequency of bone density scans a patient requires.